CLINICAL TRIAL: NCT02850107
Title: The REALITY Study: DiRectional AthErectomy + Drug-CoAted BaLloon to Treat Long, CalcifIed FemoropopliTeal ArterY Lesions
Brief Title: DiRectional AthErectomy + Drug CoAted BaLloon to Treat Long, CalcifIed FemoropopliTeal ArterY Lesions
Acronym: REALITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VIVA Physicians (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIVA-CLIN-2016-01
Record Dates: First submitted 2016-07-26; First posted 2016-07-29 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Peripheral Vascular Disease
Keywords: Atherectomy, Drug-Coated Balloon
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Non-randomized (Other): Directional Atherectomy + Drug Coated Balloon: DA followed by DCB will be performed in all enrolled subjects.
  DA includes the use of Intervention 'Medtronic HawkOne® or TurboHawk™.
  Medtronic Spider™ Distal Protection Device (DPD) is recommended for use according to IFU.
  Medtronic IN.PACT® Admiral® DCB will be used after DA.
  Volcano Visions® PV .014" IVUS catheter required to assess lesion in each procedure.
  Nitinol Stent Placement: Only FDA approved nitinol stents can be used if provisional stenting is required.
  Interventions: Device: Medtronic HawkOne® or TurboHawk™; Device: Medtronic IN.PACT® Admiral® DCB; Device: Medtronic Spider™ Distal Protection Device (DPD); Device: Volcano Visions® PV .014" IVUS catheter; Device: Nitinol Stent Placement

INTERVENTIONS:
Device: Medtronic HawkOne® or TurboHawk™ — Use of FDA Cleared Directional Atherectomy (DA) Devices. Medtronic HawkOne® Directional Atherectomy System or TurboHawk™ Plaque Excision System. DA followed by DCB will be performed in all enrolled subjects.
Device: Medtronic IN.PACT® Admiral® DCB — FDA Approved Drug Coated Balloon (DCB) Technology. Medtronic IN.PACT® Admiral® DCB will be used after DA.
Device: Medtronic Spider™ Distal Protection Device (DPD) — It is recommended that the Medtronic Spider™ Distal protection device (DPD) be paired with DA when used in complex, calcified lesions (TurboHawk™ IFU).
Device: Volcano Visions® PV .014" IVUS catheter — Lesion IVUS assessment using the Volcano Visions® PV .014" IVUS catheter will be required in all cases.
Device: Nitinol Stent Placement — Only FDA approved nitinol stents can be used if provisional stenting is required.

SUMMARY:
This study is designed to collect information during a procedure that is routine care for treating a blockage in a blood vessel in the upper part of the participant's leg. This study is for data collection reasons to help doctors gain better understanding of the treatment of disease in the blood vessels of the legs. You will be treated with two devices that are routine, or standard of care, for your doctor to treat blockages in the blood vessel of the leg. The treatment is for a blockage or narrowing caused by plaque build-up in the blood vessel. Data will be collected to assess what length of time the blood vessel will be prevented from re-narrowing through twenty-four (24) months after the procedure.

DETAILED DESCRIPTION:
This prospective study will evaluate the safety and effectiveness of two FDA 510(k) cleared DA products (Medtronic HawkOne® and TurboHawkM)19-21 and FDA approved drug-coated balloon (Medtronic IN.PACT® Admiral®)22 used in combination to debulk moderate and severely calcified femoropopliteal artery atherosclerotic lesions as defined by the published Peripheral Arterial Calcium Scoring System (PACSS) followed by treatment with the Medtronic IN.PACT® Admiral® DCB for the prevention of restenosis as assessed at 12-month follow-up. The data will be independently adjudicated by an angiographic and DUS core labs. An independent IVUS core lab to determine change in maximal luminal plaque area, pre- and post-atherectomy and post-adjunctive DCB therapy will adjudicate the assessment of debulking effectiveness. The operator will be blinded to all IVUS images and procedural success will be based on usual and customary angiographic visual assessments. The post-atherectomy plaque debulking effectiveness (change in plaque area) and vascular calcium severity as assessed by IVUS will be correlated with the angiographic metrics of RVD, pre- and post-treatment MLD, calcium grade (using PACSS), lesion length, sub-intimal wire passage, CTO length, and angiographic patterns of restenosis in all patients who sustain a CD-TLR through 12-months. All atherectomy specimens will be collected and provided to an independent histology laboratory for analysis of calcium content and vessel wall elements. The amount of embolic debris captured in the Spider® Distal Protection Device will be visually assessed. The study will validate PACSS definitions of moderate and severe calcium and its location (intimal, medial or mixed) as they relate to intra-procedural and Major Adverse Events (MAEs) through 30-day clinical follow-up (e.g., grade D-F dissections requiring provisional stenting, vessel perforation requiring an additional intervention or surgery, vessel thrombosis requiring adjunctive technologies and/or lytic agents, unplanned amputation, intra-procedure distal embolization, and CD-TLR).

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

1. Willing and able to provide informed consent;
2. Age ≥ 18 years of age;
3. Clinical evaluation determines Rutherford Category 2-4;
4. Willing to comply with all study requirements;
5. All lab work is within acceptable limits to undergo a percutaneous interventional procedure.
6. Life expectancy, in the investigator's opinion, of at least 24 months.

Angiographic Inclusion Criteria:

1. RVD ≥ 4mm and ≤ 7mm;
2. Evidence of a ≥70% de novo or restenotic lesion or occlusion in the target lesion defined as in the superficial femoral artery and/or popliteal artery, located in the arterial segment starting at least 1 cm beyond the Common Femoral Artery (CFA) bifurcation between the superficial and profunda femoris arteries (proximal anatomical landmark) to the distal P2 segment of the popliteal artery;
3. Total lesion/occlusion length:

   a. ≥ 8 cm and ≤ 18 cm
4. Total occlusion length

   a. ≥ 6 cm and ≤10 cm
5. Stenosis or occlusion begins 1cm below the profunda-SFA bifurcation;
6. Femoral or popliteal stenosis or occlusion that does not extend beyond the P2 popliteal segment;
7. Minimum 1 patent infrapopliteal vessel to the foot with ≤ 50% diameter stenosis;
8. Grade 3 or 4 intimal, medial and/or mixed calcification per the PACSS as judged by the operator at the time of the procedure;
9. Index lesion fits within guidelines below:

   9.1 If two lesions are ≤ 3 cm apart, treatment would be allowed as a single lesion providing they contain a segment of moderate or severe calcification and the total lesion length is ≥ 8 cm and ≤18 cm.

   9.2 If more than one lesion is within the target vessel, and they are separated by > 3 cm of normal vessel, one lesion must be designated by the investigator as the target lesion as long as the lesion meets all angiographic eligibility criteria. Only one index lesion is permitted for analysis, but study will allow a second lesion to be treated as a non-target lesion.
10. Infrapopliteal lesion, if diagnosed, can be staged and treated > 30 days after index procedure.

Exclusion Criteria:

General Exclusion Criteria:

1. Renal failure or chronic kidney disease with GFR ≤30 ml/min or MDRD GFR ≤30 ml/min per 1.73m2 (and serum creatinine ≥2.5 mg/dL within 30 days of index procedure);
2. Physician does not believe subject is an appropriate candidate for study;
3. Previous infra-inguinal intervention in the index limb within 30 days of the planned femoropopliteal intervention

Angiographic Exclusion Criteria:

1. Inability to cross lesion/occlusion with a guidewire or re-entry device;
2. Inability for the guidewire to re-enter and/or remain in the true lumen prior to enrollment;
3. In-stent restenosis of the target lesion, or recognition of any stent (patent or re-stenotic within the femoropopliteal segment of the index limb;
4. Aneurysm located in the target vessel or aneurysmal vessel;
5. Acute thrombus in the index limb prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

PRIMARY OUTCOMES:
Primary Patency | One year
  One-year primary patency (PSVR ≤2.4) and freedom from CD-TLR in subjects with long, moderate and severely calcified symptomatic femoropopliteal arterial stenoses and occlusions after treatment with DA+DCB.
Freedom from MAE | One month
  Freedom from (MAEs) defined as freedom from flow-limiting dissections (D-F), vessel perforations, unplanned amputation, intra-procedure distal athero-embolization and clinically-driven TVR in subjects with long, moderate and severely calcified femoropopliteal lesions and occlusions through 30 day follow up.

SECONDARY OUTCOMES:
Device Success | Post Index Procedure
  Device Success: ≤ 30% residual stenosis after completion of directional atherectomy procedure (stand-alone) as assessed by the angiographic core lab.
Procedural Success | Post Index Procedure
  Procedural Success: ≤30% residual stenosis after completion of the directional atherectomy procedure and DCB as assessed by the angiographic core lab.
IVUS | Post Index Procedure
  Core lab assessed correlation between IVUS metrics of luminal diameter, change in plaque area and luminal gain pre- and post-atherectomy, and angiographic core lab assessment of pre- and post-percent diameter stenosis (%DS) and the extent of vascular calcification will be determined
PACCS scoring and related procedural complications | 1 month
  The association of moderate and severe calcification as defined by the Peripheral Arterial Calcium Scoring System (PACSS) and the change in %DS, procedure related complications (residual stenosis ≥50%, vessel recoil and/or high-grade dissections requiring use of adjunct technologies) visual quantification of embolic material in the distal protection device and MAEs through 30-days will be assessed
Directional Atherectomy | Post Index Procedure
  Directional Atherectomy device specific metrics of total directional atherectomy time as a function of lesion length, lesion morphology, and total procedure time.
Major Adverse Events thru 24 months | 24 months
  Major adverse events through 24-months defined as composite clinically-driven target lesion revascularization (CD-TVR) defined as any re-intervention within the target vessel due to symptoms associated with a drop from post-intervention ABI/TBI >20% or >0.15, major unplanned amputation of the treated limb, and all-cause mortality post 30 day follow up through 2 year follow up.
Post procedure TVR | 6, 12, 24 months
  TVR within 6, 12, 24 months post index procedure
CD-TLR post procedure | 6, 12, 24 months
  TLR within 6, 12, 24 months post index procedure
Time to CD-TLR thru 24 months post procedure | 24 months
  Time to first clinically-driven target lesion revascularization (TLR) through 24 months post-index procedure
Major target limb amputation post procedure | 6, 12, 24 months
  Major target limb amputation within 6, 12, 24 months post index procedure
Thrombosis- target lesion post procedure | 6, 12, 24 months
  Thrombosis at the target lesion site within 6, 12, 24 months post index procedure
Primary sustained clinical improvement | 6, 12, 24 months
  Primary sustained clinical improvement: An improvement shift in the Rutherford classification of at least one class in amputation- and TVR-free surviving subjects at 6, 12, 24 months post procedure
Secondary sustained clinical improvement | 6, 12, 24 months
  Secondary sustained clinical improvement: An improvement shift in the Rutherford classification of at least one class including the need for clinically-driven TVR in amputation-free surviving subjects at 6, 12, 24 months post index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Krishna Singh, MD, Principal Investigator — VIVA Physicians, Inc.
Locations (7):
- United States (7):
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - St. Elizabeth's, Boston, Massachusetts
  - University of Mississippi, Jackson, Mississippi
  - Mount Sinai, New York, New York
  - Rex, Raleigh, North Carolina
  - Austin Heart, Austin, Texas
  - Longview Cardiac and Vascular Consultants, Longview, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Golomb BA, Dang TT, Criqui MH. Peripheral arterial disease: morbidity and mortality implications. Circulation. 2006 Aug 15;114(7):688-99. doi: 10.1161/CIRCULATIONAHA.105.593442. No abstract available. PMID 16908785
- [Result] Norgren L, Hiatt WR, Dormandy JA, Nehler MR, Harris KA, Fowkes FG, Rutherford RB; TASC II Working Group. Inter-society consensus for the management of peripheral arterial disease. Int Angiol. 2007 Jun;26(2):81-157. No abstract available. PMID 17489079
- [Result] Goodney PP, Travis LL, Nallamothu BK, Holman K, Suckow B, Henke PK, Lucas FL, Goodman DC, Birkmeyer JD, Fisher ES. Variation in the use of lower extremity vascular procedures for critical limb ischemia. Circ Cardiovasc Qual Outcomes. 2012 Jan;5(1):94-102. doi: 10.1161/CIRCOUTCOMES.111.962233. Epub 2011 Dec 6. PMID 22147886
- [Result] McKinsey JF, Zeller T, Rocha-Singh KJ, Jaff MR, Garcia LA; DEFINITIVE LE Investigators. Lower extremity revascularization using directional atherectomy: 12-month prospective results of the DEFINITIVE LE study. JACC Cardiovasc Interv. 2014 Aug;7(8):923-33. doi: 10.1016/j.jcin.2014.05.006. PMID 25147039
- [Result] Roberts D, Niazi K, Miller W, Krishnan P, Gammon R, Schreiber T, Shammas NW, Clair D; DEFINITIVE Ca(+)(+) Investigators. Effective endovascular treatment of calcified femoropopliteal disease with directional atherectomy and distal embolic protection: final results of the DEFINITIVE Ca(+)(+) trial. Catheter Cardiovasc Interv. 2014 Aug 1;84(2):236-44. doi: 10.1002/ccd.25384. Epub 2014 Feb 5. PMID 24402764
- [Result] Yazdani SK, Pacheco E, Nakano M, Otsuka F, Naisbitt S, Kolodgie FD, Ladich E, Rousselle S, Virmani R. Vascular, downstream, and pharmacokinetic responses to treatment with a low dose drug-coated balloon in a swine femoral artery model. Catheter Cardiovasc Interv. 2014 Jan 1;83(1):132-40. doi: 10.1002/ccd.24995. Epub 2013 Jul 3. PMID 23703778
- [Result] Rosenfield K, Jaff MR, White CJ, Rocha-Singh K, Mena-Hurtado C, Metzger DC, Brodmann M, Pilger E, Zeller T, Krishnan P, Gammon R, Muller-Hulsbeck S, Nehler MR, Benenati JF, Scheinert D; LEVANT 2 Investigators. Trial of a Paclitaxel-Coated Balloon for Femoropopliteal Artery Disease. N Engl J Med. 2015 Jul 9;373(2):145-53. doi: 10.1056/NEJMoa1406235. Epub 2015 Jun 24. PMID 26106946
- [Result] Tepe G, Laird J, Schneider P, Brodmann M, Krishnan P, Micari A, Metzger C, Scheinert D, Zeller T, Cohen DJ, Snead DB, Alexander B, Landini M, Jaff MR; IN.PACT SFA Trial Investigators. Drug-coated balloon versus standard percutaneous transluminal angioplasty for the treatment of superficial femoral and popliteal peripheral artery disease: 12-month results from the IN.PACT SFA randomized trial. Circulation. 2015 Feb 3;131(5):495-502. doi: 10.1161/CIRCULATIONAHA.114.011004. Epub 2014 Dec 3. PMID 25472980
- [Result] Laird JR, Schneider PA, Tepe G, Brodmann M, Zeller T, Metzger C, Krishnan P, Scheinert D, Micari A, Cohen DJ, Wang H, Hasenbank MS, Jaff MR; IN.PACT SFA Trial Investigators. Durability of Treatment Effect Using a Drug-Coated Balloon for Femoropopliteal Lesions: 24-Month Results of IN.PACT SFA. J Am Coll Cardiol. 2015 Dec 1;66(21):2329-2338. doi: 10.1016/j.jacc.2015.09.063. Epub 2015 Oct 14. PMID 26476467
- [Result] Tepe G, Zeller T, Albrecht T, Heller S, Schwarzwalder U, Beregi JP, Claussen CD, Oldenburg A, Scheller B, Speck U. Local delivery of paclitaxel to inhibit restenosis during angioplasty of the leg. N Engl J Med. 2008 Feb 14;358(7):689-99. doi: 10.1056/NEJMoa0706356. PMID 18272892
- [Result] Werk M, Langner S, Reinkensmeier B, Boettcher HF, Tepe G, Dietz U, Hosten N, Hamm B, Speck U, Ricke J. Inhibition of restenosis in femoropopliteal arteries: paclitaxel-coated versus uncoated balloon: femoral paclitaxel randomized pilot trial. Circulation. 2008 Sep 23;118(13):1358-65. doi: 10.1161/CIRCULATIONAHA.107.735985. Epub 2008 Sep 8. PMID 18779447
- [Result] Werk M, Albrecht T, Meyer DR, Ahmed MN, Behne A, Dietz U, Eschenbach G, Hartmann H, Lange C, Schnorr B, Stiepani H, Zoccai GB, Hanninen EL. Paclitaxel-coated balloons reduce restenosis after femoro-popliteal angioplasty: evidence from the randomized PACIFIER trial. Circ Cardiovasc Interv. 2012 Dec;5(6):831-40. doi: 10.1161/CIRCINTERVENTIONS.112.971630. Epub 2012 Nov 27. PMID 23192918
- [Result] Scheinert D, Duda S, Zeller T, Krankenberg H, Ricke J, Bosiers M, Tepe G, Naisbitt S, Rosenfield K. The LEVANT I (Lutonix paclitaxel-coated balloon for the prevention of femoropopliteal restenosis) trial for femoropopliteal revascularization: first-in-human randomized trial of low-dose drug-coated balloon versus uncoated balloon angioplasty. JACC Cardiovasc Interv. 2014 Jan;7(1):10-9. doi: 10.1016/j.jcin.2013.05.022. PMID 24456716
- [Result] Fanelli F, Cannavale A, Gazzetti M, Lucatelli P, Wlderk A, Cirelli C, d'Adamo A, Salvatori FM. Calcium burden assessment and impact on drug-eluting balloons in peripheral arterial disease. Cardiovasc Intervent Radiol. 2014 Aug;37(4):898-907. doi: 10.1007/s00270-014-0904-3. Epub 2014 May 9. PMID 24806955
- [Result] Rocha-Singh KJ, Zeller T, Jaff MR. Peripheral arterial calcification: prevalence, mechanism, detection, and clinical implications. Catheter Cardiovasc Interv. 2014 May 1;83(6):E212-20. doi: 10.1002/ccd.25387. Epub 2014 Feb 10. PMID 24402839
- [Result] Tepe G, Beschorner U, Ruether C, Fischer I, Pfaffinger P, Noory E, Zeller T. Drug-Eluting Balloon Therapy for Femoropopliteal Occlusive Disease: Predictors of Outcome With a Special Emphasis on Calcium. J Endovasc Ther. 2015 Oct;22(5):727-33. doi: 10.1177/1526602815600156. Epub 2015 Aug 6. PMID 26250747
- [Result] Cioppa A, Stabile E, Popusoi G, Salemme L, Cota L, Pucciarelli A, Ambrosini V, Sorropago G, Tesorio T, Agresta A, Biamino G, Rubino P. Combined treatment of heavy calcified femoro-popliteal lesions using directional atherectomy and a paclitaxel coated balloon: One-year single centre clinical results. Cardiovasc Revasc Med. 2012 Jul-Aug;13(4):219-23. doi: 10.1016/j.carrev.2012.04.007. Epub 2012 May 25. PMID 22632996
- [Derived] Rocha-Singh KJ, Sachar R, DeRubertis BG, Nolte-Ernsting CCA, Winscott JG, Krishnan P, Scott EC, Garcia LA, Baeriswyl JL, Ansel G, Rosenfield K, Zeller T; REALITY Investigators. Directional atherectomy before paclitaxel coated balloon angioplasty in complex femoropopliteal disease: The VIVA REALITY study. Catheter Cardiovasc Interv. 2021 Sep;98(3):549-558. doi: 10.1002/ccd.29777. Epub 2021 Jun 3. PMID 34080792
- See also: HawkOne 510(k) clearance. — http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfpmn/pmn.cfm?ID=K141801
- See also: Turbo Hawk 3 510(k) clearances. — http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfpmn/pmn.cfm